CLINICAL TRIAL: NCT01867580
Title: A Prospective, Randomized, Multi-Center Trial Evaluating the Effectiveness of the V.A.C. Ulta Negative Pressure Wound Therapy System With V.A.C. VeraFlo Dressing System in Operatively Debrided Wounds
Brief Title: A Pilot RCT of Veraflo With Prontosan vs VAC in Wounds Requiring Operative Debridement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: KCI USA, Inc (Industry)
Responsible Party: Sponsor
Organization: Solventum US LLC (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AHS.2011.ULTA.04
Record Dates: First submitted 2013-05-09; First posted 2013-06-04 (Estimated); Results first posted 2017-11-29 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2024-11

CONDITIONS: Wounds and Injuries
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- V.A.C.Ulta with Prontosan instillation (Experimental): Treatment Arm
  Interventions: Device: V.A.C.Ulta with Prontosan instillation
- V.A.C.Ulta without instillation (Active Comparator): Control Arm
  Interventions: Device: V.A.C.Ulta without instillation

INTERVENTIONS:
Device: V.A.C.Ulta with Prontosan instillation — NPWT with instillation of a wound cleanser (Prontosan® Wound Irrigation Solution)
  Arms: V.A.C.Ulta with Prontosan instillation
Device: V.A.C.Ulta without instillation — NPWT only
  Arms: V.A.C.Ulta without instillation

SUMMARY:
The purpose of this study is to examine the effectiveness of the Veraflo with Prontosan vs VAC in wounds that require operative debridement.

ELIGIBILITY:
Inclusion Criteria:

The Subject:

* has a wound prior to informed consent
* will be admitted as an inpatient
* is >= 18 years of age at time of consent
* is able to provide his/her own informed consent
* is willing and able to return for all scheduled and required study visits
* has an open wound >= 4cm in any plane of measurement excluding tunnels after initial surgical debridement
* has a wound that is appropriate for NPWT according to approved indications for use
* has not participated in a clinical trial within the past 30 days
* has a 30 day wound history available if the wound has been previously treated

Exclusion Criteria:

The Subject:

* is pregnant as determined by a positive serum or urine pregnancy test at the time of screening
* has a life expectancy of < 12 months
* is not healthy enough to undergo surgery for any reason
* has, in the investigator's opinion, any clinically significant condition that would impair the participant's ability to comply with the study procedures
* has, in the opinion of the investigator, a condition that will not allow the subject to tolerate the therapy (e.g. painful conditions such as vasculitis)
* has rheumatoid arthritis
* has a bleeding disorder or coagulopathy
* has a wound that contains antibiotic cement or beads
* has an ischemic lower extremity wound as determined by lack of detectable pulses in the extremity or ankle-brachial pressure indices of < 0.9 with a history of diabetes, or < 0.6 if the subject is non-diabetic
* has a known allergy or hypersensitivity to V.A.C. Therapy dressing components including polyurethane or polyvinyl alcohol (drape and foam), or materials that contain acrylic adhesive (drape adhesive)
* has a known allergy or hyper sensitivity to 3M Cavilon No Sting Barrier Film or any of its components including Hexamethyldisiloxane, isooctane, acrylate terpolymer, polyphenylmethysiloxane, copolymer
* has a know allergy or hypersensitivity to Prontosan or any of its components including polyhexamethylene biguanide (PHMB), or undecylenamidopropyl betaine
* has received NPWT on the study wound within the last 30 days
* has a wound that is contraindicated with Prontosan

  a. presence of hyaline cartilage in the wound
* has a wound that is contraindicated with V.A.C. Therapy including:

  1. malignancy in the wound
  2. untreated osteomyelitis
  3. non-enteric or unexplored fistulas
  4. necrotic tissue with eschar remaining in the wound after debridement (NOTE: Once necrotic tissue or eschar is removed from the wound bed, subjects may be included)
  5. unprotected, exposed blood vessels, anastomotic sites, organs, or nerves in direct contact with foam
* use of intervening layers between the wound bed and foam
* has a wound that is contraindicated with V.A.C. VeraFlo Therapy including:

  1. Thoracic or abdominal cavities
  2. Unexplored wounds that may communicate with adjacent body cavities
* has a wound that is closed after the initial debridement

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 181 (Actual)
Dates: Start 2013-05; Primary Completion 2015-08 (Actual); Study Completion 2015-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - Medstar Georgetown University Hospital, Washington D.C., District of Columbia
  - University of Miami Miller School of Medicine, Miami, Florida
  - Northwestern University, Chicago, Illinois
  - Brigham and Women's Hospital, Boston, Massachusetts
  - St. Luke's University Hospital, Bethlehem, Pennsylvania
  - University of Pennsylvania Health System, Philadelphia, Pennsylvania
  - University of Texas Southwestern, Dallas, Texas

RESULTS

PARTICIPANT FLOW:
Groups:
- V.A.C.Ulta With Prontosan Instillation: Treatment Arm
  V.A.C.Ulta with instillation: NPWT with instillation of a wound cleanser
Period: Overall Study
Arm/Group | V.A.C.Ulta With Prontosan Instillation | V.A.C.Ulta Without Instillation
Started | 93 | 88
Completed | 65 | 64
Not Completed | 28 | 24
Not completed — Withdrawal by Subject | 2 | 3
Not completed — Physician Decision | 17 | 12
Not completed — Lost to Follow-up | 3 | 5
Not completed — Sponsor terminated study | 1 | 0
Not completed — Missed follow-up assessment | 2 | 1
Not completed — Interruption to therapy | 3 | 0
Not completed — Osteomyelitis | 0 | 1
Not completed — Continuation of therapy | 0 | 1
Not completed — Wound recurrence | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | V.A.C.Ulta With Prontosan Instillation | V.A.C.Ulta Without Instillation | Total
Number analyzed (Participants) | 93 | 88 | 181
Age, Continuous [Median (Standard Deviation); unit: years] | 53.0 (13.92) | 52.0 (14.25) | 53.0 (14.04)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 32 | 63
  Male | 62 | 56 | 118
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 20 | 14 | 34
  Not Hispanic or Latino | 73 | 74 | 147
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 34 | 34 | 68
  White | 59 | 53 | 112
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 93 | 88 | 181

OUTCOME MEASURES:

1. Primary Outcome: Number of Inpatient Operating Room Debridements
Description: Debridement in this outcome refers to surgical removal of non viable tissue performed in an operating room
Time Frame: until the wound is deemed ready for closure or coverage by the investigator up to 64 days
Population: Per-protocol population
Measure: Count of Participants; unit: Participants
Arm/Group | V.A.C.Ulta With Prontosan Instillation | V.A.C.Ulta Without Instillation
Number analyzed (Participants) | 71 | 66
Participants
  0 debridements | 9 | 13
  1 debridement | 52 | 41
  2 debridements | 5 | 10
  3 debridements | 3 | 2
  4 debridements | 2 | 0
Statistical Analysis 1: Comparison: V.A.C.Ulta With Prontosan Instillation vs V.A.C.Ulta Without Instillation; Test type: Superiority; p = 0.6770, Regression, Logistic

2. Secondary Outcome: The Difference in Total Bacterial Counts Measured in Colony Forming Units (CFU) as Determined by Quantitative PCR Analysis.
Time Frame: Immediately following initial post debridement to the first dressing change up to 72 hours
Population: Per-protocol population (some subjects had missing assessments)
Measure: Mean (Standard Deviation); unit: Total Bacterial Counts (Log10 CFU)
Arm/Group | V.A.C.Ulta With Prontosan Instillation | V.A.C.Ulta Without Instillation
Number analyzed (Participants) | 69 | 63
Total Bacterial Counts (Log10 CFU) | -0.18 (2.15) | 0.6 (2.01)
Statistical Analysis 1: Comparison: V.A.C.Ulta With Prontosan Instillation vs V.A.C.Ulta Without Instillation; Test type: Superiority; p = 0.0202, Wilcoxon (Mann-Whitney)

3. Post Hoc Outcome: Number of Inpatient Operating Room Debridements in Surgically Dehisced Wounds
Time Frame: until the wound is deemed ready for closure or coverage by the investigator up to 64 days
Population: This only included those patients with wound etiology of Surgically Dehisced Wounds
Measure: Count of Participants; unit: Participants
Arm/Group | V.A.C.Ulta With Prontosan Instillation | V.A.C.Ulta Without Instillation
Number analyzed (Participants) | 10 | 9
Participants
  0 debridements | 3 | 1
  1 debridement | 7 | 2
  2 debridements | 0 | 4
  3 debridements | 0 | 2
  4 debridements | 0 | 0
Statistical Analysis 1: Comparison: V.A.C.Ulta With Prontosan Instillation vs V.A.C.Ulta Without Instillation; Test type: Superiority; p = 0.0142, Regression, Logistic

ADVERSE EVENTS:
Arm/Group | V.A.C.Ulta With Prontosan Instillation | V.A.C.Ulta Without Instillation
All-Cause Mortality (participants affected / at risk) | 3/93 | 1/88
Serious Adverse Events (participants affected / at risk) | 19/93 | 22/88
Other Adverse Events (participants affected / at risk) | 58/93 | 44/88
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | V.A.C.Ulta With Prontosan Instillation (N=93) | V.A.C.Ulta Without Instillation (N=88)
Osteomyelitis (Infections and infestations) | 2 | 3
Wound infection (Infections and infestations) | 1 | 3
Cellulitis (Infections and infestations) | 1 | 2
Sepsis (Infections and infestations) | 2 | 0
Abscess (Infections and infestations) | 1 | 0
Diabetic Foot Infection (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0
Purulent Discharge (Infections and infestations) | 1 | 0
Wound infection Staphylococcal (Infections and infestations) | 1 | 1
Staphylococcal infection (Infections and infestations) | 0 | 1
Wound sepsis (Infections and infestations) | 0 | 1
Transplant Failure (Injury, poisoning and procedural complications) | 3 | 2
Wound Dehiscence (Injury, poisoning and procedural complications) | 2 | 3
Wound complication (Injury, poisoning and procedural complications) | 0 | 4
Post Porcedural Haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Failure of Implant (Injury, poisoning and procedural complications) | 0 | 1
Phlebothrombosis (Vascular disorders) | 1 | 1
Wound Haemorrhage (Vascular disorders) | 1 | 1
Ischaemia (Vascular disorders) | 0 | 2
Hypotension (Vascular disorders) | 1 | 0
Peripheral Occlusive Disease (Vascular disorders) | 1 | 0
Haematoma (Vascular disorders) | 0 | 1
Aphasia (Nervous system disorders) | 1 | 0
Encephalopathy (Nervous system disorders) | 1 | 0
Grand Mal Convulsion (Nervous system disorders) | 0 | 1
Major Depression (Psychiatric disorders) | 1 | 0
Mental Status Changes (Psychiatric disorders) | 1 | 0
Aggression (Psychiatric disorders) | 0 | 1
Drug Dependence (Psychiatric disorders) | 0 | 1
Cardiac Arrest (Cardiac disorders) | 1 | 0
Cardiac Failure Congestive (Cardiac disorders) | 0 | 1
Myocardial Infarction (Cardiac disorders) | 0 | 1
Peritonitis (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Enteritis (Gastrointestinal disorders) | 0 | 1
Amputation (Surgical and medical procedures) | 1 | 0
Foot amputation (Surgical and medical procedures) | 0 | 1
Blood Glucose Fluctation (Investigations) | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1
Drug Hypersensitivity (Immune system disorders) | 0 | 1
Pneumonia Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Skin Graft Failure (Skin and subcutaneous tissue disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | V.A.C.Ulta With Prontosan Instillation (N=93) | V.A.C.Ulta Without Instillation (N=88)
Wound Dehiscence (Injury, poisoning and procedural complications) | 26 | 15
Wound Complication (Injury, poisoning and procedural complications) | 10 | 7
Skin Maceration (Skin and subcutaneous tissue disorders) | 30 | 17
Oedema (General disorders) | 14 | 8
Pain (General disorders) | 6 | 3
Glycosylated Haemoglobin Increased (Investigations) | 4 | 5
White Blood Cell Count Increased (Investigations) | 5 | 2
Constipation (Gastrointestinal disorders) | 1 | 7

LIMITATIONS AND CAVEATS:
Prontosan was used for instillation in this study. Approximately ~75% of wounds were not infected. Therefore benefits from a solution with antiseptic properties would be expected to be limited. Acelity is planning to conduct a study using saline.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less